CLINICAL TRIAL: NCT06800547
Title: Latissimus Dorsi Flap Reconstructions: Retrospective Study
Acronym: PLAST-LD
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PLAST-LD
Record Dates: First submitted 2025-01-09; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Various options for reconstruction alternatives to LD are described, as are the possible early and late side effects of LD harvesting. Currently, the choice of whether or not to resort to LD harvesting to repair the defect is based on the experience and preference of the specific working group. The importance of the study lies in the attempt to analyze the choices made in the diagnostic and therapeutic phase (demolitive and reconstructive) on patients in order to correlate the outcomes obtained in terms of healing, quality of life and complications in the recipient site and in the donor site.

DETAILED DESCRIPTION:
Currently, there are no universally accepted guidelines regarding when it is advisable to resort to a LD flap for the repair of a large defect and when it is considered contraindicated. Various options for reconstruction alternatives to LD are described, as are the possible early and late side effects of LD harvesting. Currently, the choice of whether or not to resort to LD harvesting to repair the defect is based on the experience and preference of the specific working group. The importance of the study lies in the attempt to analyze the choices made in the diagnostic and therapeutic phase (demolitive and reconstructive) on patients treated at IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola in past years, in order to correlate the outcomes obtained in terms of healing, quality of life and complications in the recipient site and in the donor site with the baseline conditions of the patients, the site and the extension of the defect.

ELIGIBILITY:
Inclusion Criteria:

* Duration of surgery, expressed in minutes;
* Hospitalization time, expressed in days;
* Need for reoperation within 30 days of the first operation;
* Survival and recurrences, based on the last available follow-up

Exclusion Criteria:

* Incomplete or missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have already undergone reconstruction surgery with a LD flap at the following U.O. Maxillofacial Surgery, Thoracic Surgery, Cardiac Surgery, Orthopedics, Urology, General Surgery, with involvement of the U.O. Plastic Surgery, from 1 January 2010 to 31 January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Technical Success | From the first enrollment, up to the 200th, an average of 2 years
  Technical success is assessed by: the duration of surgery; days of Hospitalization; need for reoperation within 30 days of the first operation; survival and recurrences, based on the last available follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pignatti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Italy